CLINICAL TRIAL: NCT05463055
Title: Varian ProBeam Proton Therapy System China Clinical Trial (Hefei)
Acronym: ProBeam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2021-03
Record Dates: First submitted 2021-12-21; First posted 2022-07-18 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Tumor, Solid
Keywords: Proton therapy; Radiation therapy; Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: a clinical study of prospective, single-arm objective performance criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm objective performance criteria (Experimental): According to the National Medical Products Administration (NMPA) Guidance on Proton and Carbon Ion treatment system clinical evaluation and clinical trial, the participants with disease control should be at least 95%. The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE grade 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  Interventions: Radiation: Proton Therapy System (ProBeam)

INTERVENTIONS:
Radiation: Proton Therapy System (ProBeam) — All of subjects (tumor patients, including tumors of the nervous system, head and neck, chest, abdomen, spine, pelvic cavity, limbs and other tumors) will be treated with Proton radiation therapy using the medical device Varian ProBeam Proton Therapy System (ProBeam). The screening period from informed consent to enrollment is expected to be 4 weeks, while the treatment period is 1 to 8 weeks. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up will be 3 months after the end of the last treatment. Total expected participation for each subject from screening to the completion of short-term follow-up is a maximum duration of 12 weeks + 3 months ( for this trial). Long-term follow-up continues after the end of short-term follow-up until the 5th year after the end of the last radiotherapy session.

SUMMARY:
This study is prospective, two-center, single-arm objective performance criteria. This trial will be conducted in 2 clinical trial sites with a total of 47 subjects enrolled. All of subjects will be treated with radiation therapy using the medical device Varian ProBeam Proton Therapy System (ProBeam), aim to compare the data with objective performance criteria to evaluate the effectiveness and safety of ProBeam radiotherapy system for oncology patients, providing clinical evidence for the medical device registration.

DETAILED DESCRIPTION:
Oncology patients, including tumors of the nervous system, head and neck, chest, abdomen, spine, pelvic cavity, limbs and other tumors. The screening period from informed consent to enrollment is expected to be 4 weeks, while the treatment period is 1 to 8 weeks. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months after treatment completion and long-term follow-up is 5 years after the end of the last radiotherapy session.

The clinical trial with short-term follow-up fulfills the requirements for National Medical Products Administration (NMPA) regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.

Long-term follow-up report will be submitted for future post market evaluation when requested by NMPA.

ELIGIBILITY:
Inclusion Criteria (Major Criteria):

1. 18≤ age≤ 80 years;
2. First-diagnosed patients with tumors of the nervous system, head and neck, chest, abdomen, spine, pelvic cavity, limbs, etc. by tissue/cell pathology;
3. Eastern Cooperative Oncology Group (ECOG) physical condition is graded as 0 to 2;
4. Women of childbearing had negative results in the blood pregnancy test (Human Chorionic Gonadotropin, HCG) 7 days prior to the first treatment;
5. The subject or subject's guardian is able to understand the purpose of the study, demonstrate sufficient compliance with the protocol and sign informed consent form.

Exclusion Criteria (Major Criteria):

1. The subject with radiotherapy contraindications, including the known genetic tendencies that increase the sensitivity of normal tissue radiotherapy or the accompanying diseases that lead to hypersensitivity to radiotherapy;
2. The subject with other uncontrolled tumors except that to be treated according to medical history or the investigator's estimation, or with other malignant tumors within five years prior to enrollment;
3. Implanted pacemakers or other metal prosthesis within the scope of proton therapy;
4. Other situations that investigator determines not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-12-26 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Zhang, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from December 2021 to June 2022. The location of the study was in medical clinic.
Pre-assignment Details: Subjects meeting the inclusion/exclusion criteria and enrolled in the trial were treated with ProBeam Proton Therapy System (ProBeam) unless the subject's status isn't fit for proton therapy prior to treatment during treatment planning and target area confirming. For example, if the subject's treatment plan indicated that within the target area wasn't suitable for radiation therapy, then should preclude from the trial.
Groups:
- Single-arm Objective Performance Criteria: The primary effectiveness for clinical trial should be 95% participants with disease control, which includes Complete Response, Partial Response and Stable Disease. The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE level 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  Participants enrolled will be treated with Proton radiation therapy. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months and long-term follow-up is 5 years after treatment completion.
  The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by National Medical Products Administration (NMPA). Therefore, long-term follow-up result will not be reported here.
Period: Overall Study
Arm/Group | Single-arm Objective Performance Criteria
Started | 47
Completed | 45
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Single-arm Objective Performance Criteria: The primary effectiveness for clinical trial should be 95% participants with disease control, which includes Complete Response, Partial Response and Stable Disease. The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE level 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  All enrolled subjects were treated with ProBeam Proton Therapy System. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months after treatment completion and long-term follow-up is 5 years after treatment completion. The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by NMPA. Therefore, long-term follow-up result will not reported here.
Arm/Group | Single-arm Objective Performance Criteria
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han of Chinese | 47
single-arm objective performance criteria [Count of Participants; unit: Participants] | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Control
Description: Disease control refers to partial response and stable disease and complete response. Percentage of participants with disease control should be at least 95%.
  Tumor disease control measured by Magnetic Resonance Imaging (MRI)/Computed Tomography (CT) using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). CT or MRI changes will be assessed before and after treatment.
Time Frame: 3 months ± 7 days after treatment completion, up to 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Single-arm Objective Performance Criteria: The primary effectiveness for clinical trial should be 95% participants with disease control, which includes Complete Response, Partial Response and Stable Disease. The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE level 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  Subjects enrolled in the trial will be treated with Proton radiation therapy. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months and long-term follow-up is 5 years after treatment completion.
  The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by National Medical Products Administration (NMPA). Therefore, long-term follow-up result will not be reported here.
Arm/Group | Single-arm Objective Performance Criteria
Number analyzed (Participants) | 45
percentage | 100 [92.1 to 100]

2. Primary Outcome: Percentage of Participants With Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 Toxic Reaction
Description: The percentage of participants with CTCAE grade 3 toxic reaction should be lower than 5%. Higher than 5% means worse outcome and will not be accepted.
  AEs occurred in the clinical trial are recorded and scored by the investigator according to CTCAE version 5.0.
Time Frame: From enrollment to 3 months ± 7 days after treatment completion, up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Single-arm Objective Performance Criteria: The primary effectiveness for clinical trial should be 95% participants with disease control, which includes Complete Response, Partial Response and Stable Disease. The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE level 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial use single-arm objective performance criteria.
  Subjects enrolled in the trial will be treated with Proton radiation therapy. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months and long-term follow-up is 5 years after treatment completion.
  The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by National Medical Products Administration (NMPA). Therefore, long-term follow-up result will not be reported here.
Arm/Group | Single-arm Objective Performance Criteria
Number analyzed (Participants) | 47
Participants | 0

3. Primary Outcome: Percentage of Participants With Common Terminology Criteria for Adverse Events (CTCAE) Grade 4 and 5 Toxic Reaction
Description: The percentage of subjects with toxic reactions of levels 4 and 5 should be 0%. If CTCAE level 4 and 5 toxic reaction occured, the clinical trial is considered as failure.
  AEs occurred in the clinical trial are reported and scored by the investigator according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: From enrollment to 3 months ± 7 days after treatment completion, up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm Objective Performance Criteria
Number analyzed (Participants) | 47
Participants | 0

ADVERSE EVENTS:
Time Frame: The clinical trial started from subject enrollment to 3 months ± 7 days after the last treatment, up to 24 weeks. Long-term follow-up report (from 3-month follow-up till 5 years) will be submitted for future post market evaluation when requested by NMPA. Therefore, long-term follow-up result will not be reported here.
Groups:
- Single-arm Objective Performance Criteria: The primary effectiveness for clinical trial should be 95% participants with disease control, which includes Complete Response, Partial Response and Stable Disease. The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) level 3 toxic reaction should be lower than 5%, CTCAE level 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  Subjects enrolled in the trial will be treated with Proton radiation therapy. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months and long-term follow-up is 5 years after treatment completion.
  The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by National Medical Products Administration (NMPA). Therefore, long-term follow-up result will not be reported here.
Arm/Group | Single-arm Objective Performance Criteria
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 9/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm Objective Performance Criteria (N=47)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm Objective Performance Criteria (N=47)
Radiation dermatitis (Injury, poisoning and procedural complications) | 9 (9)
Radiation mucositis (Injury, poisoning and procedural complications) | 3 (3)
hair loss (General disorders) | 3 (3)
Low White blood cell count (Blood and lymphatic system disorders) | 2 (2)
Increased skin pigmentation (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release. Sponsor have the right to require Principal Investigator, as applicable, to remove specifically identified Confidential Information (other than Trial Data) and/or to delay the proposed publication, presentation or other public disclosure for an additional sixty (60) days to enable Sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT05463055/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT05463055/SAP_001.pdf